CLINICAL TRIAL: NCT03969394
Title: The Prognostic Role of the Right Ventricle in Patients With Heart Failure or Congenital Heart Disease
Acronym: RV-STRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/02MAR/117
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
Keywords: strain; MRI; echocardiography
MeSH Terms: conditions — Heart Failure; Sprains and Strains | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Failure Patients (Experimental): Patients with Heart Failure
  Interventions: Diagnostic Test: Medical imaging

INTERVENTIONS:
Diagnostic Test: Medical imaging — Medical Imaging consisting of 1 MRI and 1 echocardiography at baseline

SUMMARY:
The objectives are

1. to validate quantification of 2D and 3D right ventricular strian measurements of right ventricular performance in cross comparison to cardiac MRI and to evaluate its relation to right ventricular fibrosis.
2. to evaluate their prognostic value in patients with heart failure with either depressed or preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with heart failure

Exclusion Criteria:

* Renal failure
* Contraindications to Cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
Heart Failure | 3 years
  Hospitalization due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Gerber, MD,PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houard L, Amzulescu MS, Colin G, Langet H, Militaru S, Rousseau MF, Ahn SA, Vanoverschelde JJ, Pouleur AC, Gerber BL. Prognostic Value of Pulmonary Transit Time by Cardiac Magnetic Resonance on Mortality and Heart Failure Hospitalization in Patients With Advanced Heart Failure and Reduced Ejection Fraction. Circ Cardiovasc Imaging. 2021 Jan;14(1):e011680. doi: 10.1161/CIRCIMAGING.120.011680. Epub 2021 Jan 13. PMID 33438438